CLINICAL TRIAL: NCT04187742
Title: Feedback to Improve Rational Strategies of Antibiotic Initiation and Duration in Long Term Care (Phase 2)
Brief Title: Feedback to Improve Rational Strategies of Antibiotic Initiation and Duration in Long Term Care (FIRST AID -LTC) - Phase 2
Acronym: FIRST AID-LTC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for Clinical Evaluative Sciences (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Ontario Agency for Health Protection and Promotion (Other Government); Health Quality Ontario (Other)
Responsible Party: Principal Investigator, Nick Daneman, Adjunct Scientist, Institute for Clinical Evaluative Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 441-2017 (Phase 2)
Record Dates: First submitted 2019-12-03; First posted 2019-12-05 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Antibiotic Initiation; Antibiotic Duration

STUDY DESIGN:
Intervention Model Description: Assess three interventional parallel study models consisting of two intervention arms each
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The team at Health Quality Ontario will be aware of the physicians' assignment to the different email interventions so that they can send the correct audit-and-feedback report email announcements. However, the analytic team at ICES will be masked, and outcome data will be extracted by the analysis team from routinely collected administrative databases and report opening metrics that cannot be linked back to the original intervention assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- LTC Physicians Receive Social Comparison Email (Active Comparator): All LTC physicians who receive a social comparison email
  Interventions: Behavioral: Social Comparison Email vs. Standard Email
- LTC Physicians Do Not Receive Social Comparison Email (No Intervention): All LTC physicians who do not receive a social comparison email
- LTC Physicians Receive Maintenance Certification Email (Active Comparator): All LTC physicians who receive a maintenance certification email
  Interventions: Behavioral: Maintenance Certification Email vs. Standard Email
- LTC Physicians Do Not Receive Maintenance Certification Email (No Intervention): All LTC physicians who do not receive a maintenance certification email
- LTC Physician Has (or has not) Opened Prior Report (Active Comparator): LTC physicians who opened (or has not opened) at least one report receive an email informing them of their report opening status
  Interventions: Behavioral: Report Opening Status Email vs. Standard Email (among previous report openers and non-openers)
- LTC Physician Has (or has not) Opened Prior Report (Control) (No Intervention): LTC physicians who opened (or has not opened) at least one report receive a standard email without report opening status

INTERVENTIONS:
Behavioral: Social Comparison Email vs. Standard Email — Evaluate whether emails with social comparison incentives will encourage greater report opening by physicians leading to greater reductions in antibiotic use, than a standard email without social comparison incentives
  Arms: LTC Physicians Receive Social Comparison Email
Behavioral: Maintenance Certification Email vs. Standard Email — Evaluate whether emails with maintenance certification incentives will encourage greater report opening by physicians leading to greater reductions in antibiotic use, than a standard email without social comparison incentives
  Arms: LTC Physicians Receive Maintenance Certification Email
Behavioral: Report Opening Status Email vs. Standard Email (among previous report openers and non-openers) — Evaluate whether emails informing physicians of their report opening status (among those who have previously opened at least one report and those who have never opened a report) will encourage greater report opening by physicians leading to greater reductions in antibiotic use, than a standard email without report opening status information
  Arms: LTC Physician Has (or has not) Opened Prior Report

SUMMARY:
There is a high rate of inappropriate antibiotic use in LTC facilities, with both unnecessary initiation and prolongation of treatments. Although there are challenges to rational antibiotic use in LTC, the variability in antibiotic initiation and use of prolonged treatment durations is driven by prescriber tendencies rather than resident characteristics. Audit-and-feedback is a well-established intervention to improve professional practices, and is ideally suited for use to improve antibiotic prescribing tendencies in LTC. The literature is saturated with trials indicating benefit of audit-and-feedback, but is in dire need of studies to identify methods to improve the impact of this technique. Health Quality Ontario (HQO), a key partner in the FIRST AID-LTC research program, is already providing audit-and-feedback for other inappropriate prescribing practices in LTC, and has identified antibiotic prescribing as a priority focus.

DETAILED DESCRIPTION:
The overarching goals of FIRST AID - LTC are two-fold:

1. Improve rational antibiotic prescribing by physicians to minimize harms among LTC residents.
2. Advance the science of audit-and-feedback to improve physician prescribing practices.

Specific Aims

To advance audit-and-feedback implementation science:

1. by determining whether social comparison incentives, personal maintenance of certification incentives, and informing physicians of their report opening status (i.e., never opened a report vs. opened at least one report), can lead to increased opening of the feedback report and greater reductions in antibiotic use than standard email messaging.

Anticipated Contributions to Health-Related Knowledge

Although the literature is inundated with trials examining the impact of audit-and-feedback compared to usual care, there is a need for studies to improve audit-and-feedback delivery. FIRST AID-LTC will test optimal delivery and peer comparison techniques for audit-and-feedback. The knowledge learned can be extrapolated to antibiotic interventions in LTC in other provinces across Canada, as well more broadly to inappropriate medication prescribing practices in LTC.

Anticipated Contributions to Health Care, Health Systems and Health Outcomes

FIRST AID-LTC will lead to immediate reductions in excess antibiotic use in Ontario LTC facilities, which in turn should result in substantial reductions in direct drug costs, as well as downstream complications of allergy, organ toxicity, C. difficile infections and antimicrobial resistance. With easy transferability to other Canadian provinces, the improvements in cost-savings and patient outcomes could be massive in scope.

ELIGIBILITY:
To Identify an LTC Resident

Inclusion Criteria:

An individual having a minimum of 2 records on separate days within the quarter meeting any combination of the following criteria:

* a record for a non-emergency long-term care inpatient service OR
* an Ontario Drug Benefits record administered in long-term care

Index date = The analysis will be anchored on the most recent of either of the records above with a given quarter or their date of death (whichever date is earliest)

Exclusion Criteria:

* Non-Ontario resident at index date
* Invalid age (age<19 or age>115) at index date
* Missing or invalid sex or date of birth at index date
* Death date is >7 days before index date
* If the individual does not live in a nursing home or home for the aged
* Cannot be linked to a Most Responsible Physician (MRP) (see methodology below)

To identify the Most Responsible Physician (MRP) Using Virtual Rostering

For each patient in the above resident cohort, the study team will retrieve all records from health care providers in the 6 month period preceding the index date (180 days), keeping only records from physicians who have a specialty of 1) general practice, 2) community medicine or 3) geriatrics.

Steps for MRP assignment:

Step 1) The study team will first select physicians with highest count of OHIP records for the monthly management of a nursing home or home for the aged. This is completed for as many residents as possible.

Step 2) If there were no monthly management fee records as described above then the physician with the highest count of non-emergency long-term care inpatient services records for each patient will be selected. This step is only applied to residents who could not be matched to a physician by Step 1. **Physician must have seen the patient one or more times in 90 days prior to and including index date to be considered MRP. This criteria is applied to ensure the physician has seen the resident within the reporting quarter.

Step 3) Some patients will virtually roster to physicians in Enrollment groups, some will virtually roster to physicians that are not in a group. For these, we will recode enrollment program type to 'NOR' (not otherwise rostered) - these are likely fee for service physicians.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 421 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Rate of report opening | 3 months
  Percentage of physicians opening/accessing the report at least once in the 3 month interval following email send out

SECONDARY OUTCOMES:
ER visit or hospitalization for infection | 3 months
  The percentage of a LTC physicians' patients that experienced an ER visit or hospitalization due to a potential antibiotic-related harm, including: allergy, general medicine adverse event, diarrhea, C. difficile infection, or infection with an antibiotic-resistant organism
ER visit or hospitalization for antibiotic harms | 3 months
  To test for harms related to decreased antibiotic use by comparing the percentage of LTC physicians' patients that experience an infection-related ER visit or admission
Net clinical impact | 3 months
  Measure the net clinical impact of the intervention, by comparing all-cause ER visits and hospitalizations and mortality
Anti-psychotic use | 3 months
  The percent reduction in anti-psychotic use
Benzodiazepine use | 3 months
  The percent reduction in benzodiazepines
Antibiotic initiation | 3 months
  Percentage of patients initiated on an antibiotic
Antibiotic duration | 3 months
  Percentage of antibiotic treatments prolonged > 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Nick Daneman, MD, Principal Investigator — ICES
Locations (1):
- ICES, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Daneman N, Lee S, Bai H, Bell CM, Bronskill SE, Campitelli MA, Dobell G, Fu L, Garber G, Ivers N, Kumar M, Lam JMC, Langford B, Laur C, Morris AM, Mulhall CL, Pinto R, Saxena FE, Schwartz KL, Brown KA. Behavioral Nudges to Improve Audit and Feedback Report Opening Among Antibiotic Prescribers: A Randomized Controlled Trial. Open Forum Infect Dis. 2022 Mar 2;9(5):ofac111. doi: 10.1093/ofid/ofac111. eCollection 2022 May. PMID 35392461